CLINICAL TRIAL: NCT01876654
Title: Evaluation of the TruMatch® Personalized Solutions System in Knee Prosthetic Surgery
Brief Title: Evaluation of the TruMatch® System in Knee Prosthetic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Pietro Randelli, MD, Assistant Professor, University of Milan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TruMatch02
Record Dates: First submitted 2013-06-10; First posted 2013-06-12 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Osteoarthritis, Knee
Keywords: Total Knee Replacement; Patient specific instrumentation
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TruMatch® patient specific cutting guide (Experimental): In patients randomized to experimental arm, TKR components will be implanted using TruMatch® patient specific cutting guides.
  Interventions: Device: TruMatch® patient specific cutting guide
- Conventional cutting guide (No Intervention): In patients randomized to control arm, TKR components will be implanted using Attune® instrumentation (femoral intra-medullary guide, tibial extra-medullary guide), without TruMatch® patient specific cutting guides.

INTERVENTIONS:
Device: TruMatch® patient specific cutting guide
  Other Names: TruMatch® Personalized Solutions (DePuy).
  Arms: TruMatch® patient specific cutting guide

SUMMARY:
Patient specific instrumentation is an alternative to conventional intra- and extra-medullary guides to perform the femoral and tibial cuts in total knee replacement (TKR).

This instrumentation could provide a better alignment of a TKR, reduce blood losses and operative time, and improve clinical outcomes.

The primary goal of this study is to compare the femorotibial mismatch angle of two groups of patients: patients undergoing posterior stabilized, fixed bearing TKR with conventional Attune® instrumentation (DePuy Johnson & Johnson, Warsaw, Indiana), versus patient undergoing TKR with the TruMatch® (DePuy Johnson & Johnson, Warsaw, Indiana) cutting guide.

DETAILED DESCRIPTION:
Good alignment after a TKR leads to faster rehabilitation, better clinical outcomes and lower revision rate. A correct rotational (axial) alignment reduces patellofemoral complications, polyethylene wear and unexplained knee pain.

A randomized controlled study is conducted to test if to use the TruMatch® (DePuy Johnson & Johnson, Warsaw, Indiana) patient specific instrumentation reduces the number of patients presenting femorotibial mismatch.

Secondary goals are to compare:

* alignment in the coronal, sagittal and axial plane of the femoral component;
* alignment in the coronal and sagittal plane of the tibial component;
* number of recuts during surgery and surgeon's adherence to planning;
* blood loss;
* clinical outcome after two months using the Oxford Knee Score (OKS).

After having signed informed consent, patients will be randomized in 2 groups preoperatively. A long-leg CT scan, according to manufacturer's instructions, will be performed on patients randomized to the TruMatch® group.

Haemoglobin and haematocrit will be recorded pre- and postoperatively.

Two months after surgery a knee CT-scan, anteroposterior and laterolateral scanograms will be performed on all patients, and OKS will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age > 40, <80
* Indication for TKR
* Surgical indication for Attune®, posterior stabilized, fixed bearing TKR
* Patients signed written informed consent

Exclusion Criteria:

* Age > 80, < 40
* TKR revision surgery
* Metal devices within 8 cm from knee articular surfaces
* Fixed knee deformities greater than 15° in varus, valgus, flexion or tibial slope.
* Knee ankylosis
* Previous tibial osteotomy surgery
* Informed consent not accepted
* Serious comorbidity
* Active infections
* Pregnant or breastfeeding women

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Femorotibial mismatch angle | 2 months after surgery
  Angle between the posterior femoral condylar plane and the plane passing trough the posterior end of the tibial keel (measured on axial CT-scan).

SECONDARY OUTCOMES:
Knee function | 2 months after surgery
  For evaluation of knee function, patients will be asked to fill in the OKS questionnaire.

OTHER OUTCOMES:
Operative time | During surgery
  Tourniquet application time will be recorded during surgery.
Blood loss | 3-7 days after surgery
  Intra- and post-operative blood loss will be measured and compared between the two treatment arms.
Alignment | 2 months after surgery
  Coronal limb alignment, alignment in the coronal, sagittal and axial plane of the femoral component and alignment in the coronal and sagittal plane of the tibial component will be measured using a knee CT-scan, anteroposterior and laterolateral scanograms.

CONTACTS AND LOCATIONS:
Overall Officials: Pietro S. Randelli, MD, Principal Investigator — University of Milan
Locations (1):
- Unità Operativa Ortopedia II, Policlinico San Donato (Istituto di Ricovero e Cura a Carattere Scientifico), San Donato Milanese, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fang DM, Ritter MA, Davis KE. Coronal alignment in total knee arthroplasty: just how important is it? J Arthroplasty. 2009 Sep;24(6 Suppl):39-43. doi: 10.1016/j.arth.2009.04.034. Epub 2009 Jun 24. PMID 19553073
- [Background] Longstaff LM, Sloan K, Stamp N, Scaddan M, Beaver R. Good alignment after total knee arthroplasty leads to faster rehabilitation and better function. J Arthroplasty. 2009 Jun;24(4):570-8. doi: 10.1016/j.arth.2008.03.002. Epub 2008 May 19. PMID 18534396
- [Background] Nunley RM, Ellison BS, Zhu J, Ruh EL, Howell SM, Barrack RL. Do patient-specific guides improve coronal alignment in total knee arthroplasty? Clin Orthop Relat Res. 2012 Mar;470(3):895-902. doi: 10.1007/s11999-011-2222-2. Epub 2011 Dec 20. PMID 22183477
- [Background] Chauhan SK, Clark GW, Lloyd S, Scott RG, Breidahl W, Sikorski JM. Computer-assisted total knee replacement. A controlled cadaver study using a multi-parameter quantitative CT assessment of alignment (the Perth CT Protocol). J Bone Joint Surg Br. 2004 Aug;86(6):818-23. doi: 10.1302/0301-620x.86b6.15456. PMID 15330021
- [Background] Bell SW, Young P, Drury C, Smith J, Anthony I, Jones B, Blyth M, McLean A. Component rotational alignment in unexplained painful primary total knee arthroplasty. Knee. 2014 Jan;21(1):272-7. doi: 10.1016/j.knee.2012.09.011. Epub 2012 Nov 7. PMID 23140906
- [Background] Rienmuller A, Guggi T, Gruber G, Preiss S, Drobny T. The effect of femoral component rotation on the five-year outcome of cemented mobile bearing total knee arthroplasty. Int Orthop. 2012 Oct;36(10):2067-72. doi: 10.1007/s00264-012-1628-0. Epub 2012 Aug 1. PMID 22851124
- [Background] Heyse TJ, Tibesku CO. Improved femoral component rotation in TKA using patient-specific instrumentation. Knee. 2014 Jan;21(1):268-71. doi: 10.1016/j.knee.2012.10.009. Epub 2012 Nov 8. PMID 23140905
- [Derived] Randelli PS, Menon A, Pasqualotto S, Zanini B, Compagnoni R, Cucchi D. Patient-Specific Instrumentation Does Not Affect Rotational Alignment of the Femoral Component and Perioperative Blood Loss in Total Knee Arthroplasty: A Prospective, Randomized, Controlled Trial. J Arthroplasty. 2019 Jul;34(7):1374-1381.e1. doi: 10.1016/j.arth.2019.03.018. Epub 2019 Mar 13. PMID 30979672